CLINICAL TRIAL: NCT03206359
Title: Evaluation of GADD34 and Type I IFN Response Gene Expression in Patients Suffering From Systemic Lupus Erythematosus
Brief Title: GADD34 and Type I IFN Response Genes in SLE
Acronym: GADD34-IFN
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.197
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-06

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Unfolded Protein Response; GADD34; Type I IFN; IFN response genes; Type II IFN; anti-DNA autoantibodies
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with SLE
- Healthy subjects

SUMMARY:
GADD34 (Growth Arrest and DNA Damage inducible-protein) is a regulatory subunit of PP1 (phosphatase 1) phosphatase which dephosphorylates eIF2alpha (eucaryotic initiation factor 2 alpha subunit), representing a negative feedback loop of the unfolded protein response (UPR). Moreover, GADD34 is necessary for type I interferon (IFN) production in response to viral infection in murine models. We investigate here the expression of GADD34 in systemic lupus erythematosus (SLE), in which type I IFN has an important pathogenic role.

We report a case-control study on GADD34 gene expression in PBMC (peripheral blood mononuclear cells) of SLE patients (n=60) and age- and sex-matched healthy controls (n=30). The level of GADD34 gene expression, as well as of type-I IFN response genes in PBMC is measured by quantitative PCR.

ELIGIBILITY:
Inclusion Criteria:

* Man and woman over 18 years old.
* Patients suffering from SLE (SLICC criteria)
* Patients having given their "Non-opposition"
* Patients with social security affiliation (required in France)

Exclusion Criteria:

* Patients suffering from other auto-immune disease (except SAPL, thyroiditis, and Gougerot Sjogren syndrome)
* Patients with viral infection within 15 days
* People with special protection (defined in articles L1121-§5-8 and articles L3212-§1-3 of French health care law)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients suffering from systemic lupus erythematosus
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2012-01-25 (Actual); Primary Completion 2015-04-03 (Actual); Study Completion 2015-04-03 (Actual)

PRIMARY OUTCOMES:
GADD34 expression in SLE patients | 4 years
  Evaluation of GADD34 expression in PBMC of patients suffering from SLE compared to GADD34 expression in PBMC of healthy subjets. GADD34 gene expression level is quantified in the PBMC by quantitative PCR

SECONDARY OUTCOMES:
GADD34 and IFN response gene expression | 4 years
  Evaluation of the relation between IFN response gene expression and GADD34 expression in PBMC of patients suffering from SLE. IFN response gene and GADD34 expression level is quantified in the PBMC by quantitative PCR
GADD34 expression and pathology activity | 4 years
  Evaluation of the relation between GADD34 overexpression and the activity of the pathology
GADD34 expression and pathology activity | 4 years
  Evaluation of the relation between GADD34 overexpression and the presence of anti-DNA antibodies.
CHOP and BiP expression | 4 years
  Evaluation of the expression of other genes of UPR (like CHOP and BiP) in PBMC of patients with SLE, compared to the expression of these genes in PBMC of healthy subjets.

IPD SHARING:
Plan to Share IPD: No